CLINICAL TRIAL: NCT02777762
Title: Strategies to Promote Physical Activity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michaela Kiernan, Senior Research Scientist, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37737; R01HL128666 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-05-19 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fun First (Experimental): Strategies to promote enjoyment of physical activity
  Interventions: Behavioral: Fun First
- Close at Hand (Active Comparator): Strategies to promote tracking of physical activity
  Interventions: Behavioral: Close at Hand

INTERVENTIONS:
Behavioral: Fun First — 8 weekly interactive small-group sessions with a health coach
  Arms: Fun First
Behavioral: Close at Hand — 8 weekly check-ins with a state of the art, engaging mobile app
  Arms: Close at Hand

SUMMARY:
Getting regular physical activity has many health benefits. Current physical activity programs often encourage people to track their physical activity as a way to motivate them to continue being physically active over time. However, not everyone enjoys physical activity, so tracking physical activity may not be very motivating. This research study will evaluate whether a new program-specifically designed to enhance people's enjoyment of physical activity-improves people's attitudes toward physical activity compared to a program that encourages people to track their physical activity with a mobile app.

ELIGIBILITY:
Inclusion Criteria:

1. 25 ≤ BMI ≤ 39 kg/m2
2. Systolic blood pressure 120-139 mmHg and/or diastolic blood pressure 80-89 mmHg
3. Not currently taking medications for blood pressure

Exclusion Criteria:

1. Not free of diagnosed heart disease, diabetes, and cancer
2. Medical contraindications to regular, unsupervised physical activity
3. Not stable on all medications over the past 3 months
4. Not free of binge eating disorder or bulimic compensatory symptoms
5. No regular access to a mobile phone and Internet
6. Not able to speak and understand English
7. Currently pregnant or planning to be within the next year
8. Planning to move in the next year
9. Not willing to be randomized

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported enjoyment of physical activity assessed with the Behavioral Regulation in Exercise Questionnaire Version 2 (BREQ-2) Intrinsic Regulation subscale | Change from baseline to 2 months
  Survey questions

SECONDARY OUTCOMES:
Change in self-reported physical activity assessed with the Stanford Leisure-Time Categorical Item (L-Cat) | Change from baseline to 2 months
  Survey question

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Kiernan, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States